CLINICAL TRIAL: NCT02461537
Title: Evaluation of the Impact of Remission Induction Chemotherapy Prior to Allogeneic Stem Cell Transplantation in Relapsed and Poor-response Patients With AML
Brief Title: Impact of Remission Induction Chemotherapy Prior to Allogeneic SCT in Relapsed and Poor-response Patients With AML
Acronym: ETAL3-ASAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: DKMS gemeinnützige GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DKMS-14-01; 2014-003124-44 (EudraCT Number)
Record Dates: First submitted 2015-05-28; First posted 2015-06-03 (Estimated); Last update posted 2024-01-19 (Actual); Status verified 2022-08

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIST(remission induction) (Active Comparator): high-dose cytarabine 3 g/m2 (days 1-3)/mitoxantrone 10mg/m2 (days 3-5)
  Interventions: Drug: HAM
- DISC (disease control) (Experimental): low-dose cytarabine 20 mg/ m2 and /or mitoxantrone 10mg/m2
  Interventions: Drug: LDAC and/or Mitoxantrone

INTERVENTIONS:
Drug: HAM — High-dose cytarabine 1 - 3 g/m2 (days 1-3)/Mitoxantrone 20 mg/m2 (days3-5)
  Arms: RIST(remission induction)
Drug: LDAC and/or Mitoxantrone — Low-dose cytarabine 20 mg/m2 (days 1-10) and/ or mitoxantrone 10mg/m2 (max 3 doses)
  Arms: DISC (disease control)

SUMMARY:
This trial compares outcome of two treatment strategies for patients with high-risk AML who failed to achieve or maintain a complete remission with standard therapy. Patients will be randomized between two strategies. The standard strategy is aimed at achieving a complete remission by aggressive salvage chemotherapy using high dose cytarabine and mitoxantrone, . The alternative is a less toxic disease-control strategy of disease monitoring and, if necessary, low-dose cytarabine or mitoxantrone prior to allogeneic transplantation, which should be performed as soon as possible.

DETAILED DESCRIPTION:
Patients with high-risk acute myeloid leukemia (AML) who relapsed or showed a poor response to induction chemotherapy have a dismal prognosis. For these patients, allogeneic transplantation is the recommended treatment. While allogeneic transplantation may be considered as the ultimate treatment concept, the treatment path to transplantation is not well defined.

The traditional approach to pursue a complete remission by means of aggressive reinduction chemotherapy prior to allogeneic transplantation. This approach is associated with potentially life-threatening toxicities and has limited efficacy. As a result, only some patients will reach allogeneic transplantation in complete remission.

To reduce the number of patients who die or who are ineligible for transplantation due to the toxicity of aggressive induction chemotherapy, other bridging options have been explored. One promising alternative is to abstain from remission induction. Instead, disease control by means of less aggressive chemotherapy or simply monitoring leukemic proliferation can be considered.

This randomized trial will identify if there is non-inferiority of the less toxic approach, compared to the standard approach of remission induction by aggressive chemotherapy prior to allogeneic transplantation.

ELIGIBILITY:
Inclusion Criteria

* Signed written informed consent.
* Male and female patients of 18 to 75 years of age.
* Diagnosis of AML according to WHO criteria.
* Patient is fit for aggressive induction chemotherapy and transplantation by assessment of an experienced hematologist.
* No history of chronic pulmonary disease and absence of dyspnea. Otherwise, documented diffusion lung capacity for carbon monoxide ( DLCO ) ≤ 40 percent ( adjusted for hemoglobin, if available ) and FEV1 / FVC ≥ 50 percent.
* HLA - identical sibling. or
* HLA - compatible unrelated donor ( ≥ 9 /10 antigens matched for HLA - A, - B, - C, -DRB 1, and - DQB 1 ) with completed confirmatory typing or
* Two unrelated donors with > 90 percent probability of a 9 /10 match for HLA - A, - B, - C, - DRB 1, and - DRQB 1, according to Opti Match ® list.

For the relapse stratum

* First AML relapse, defined as ≥ 5 percent bone marrow blasts and / or extramedullary AML manifestation.

For the poor - responders stratum

* AML that evolves from previously documented myelodysplastic syndrome ( MDS ),

and / or

* diagnosis of therapy-related myeloid neoplasm ( t - MN ), and / or

a ) If patient ≤ 60 years old adverse risk AML according to ELN - criteria and ≥ 5 percent bone marrow blasts after the first cycle of induction therapy.

b ) If patient > 60 years old non-favourable risk AML according to ELN - criteria and ≥ 5 percent bone marrow blasts after the first cycle of induction therapy.

Exclusion Criteria

* Acute promyelocytic leukemia ( APL ).
* WBC count of ≥ 50 GPt / L at study inclusion.
* For patients in the poor - responder stratum the first cycle of induction therapy must not contain HDAC, defined as cytarabine at single-doses of > 1 g / m 2.
* Patient has received more than 440 mg / m2 daunorubicin equivalents.
* Severe organ dysfunction, defined as
* Left ventricular ejection fraction < 50 percent.
* Patients who receive supplementary continuous oxygen.
* Serum bilirubin > 1.5 x ULN ( if not considered Gilbert-Syndrome ), ASAT / ALAT > 5 x ULN.
* Estimated GFR < 50 ml / min.
* Treatment with any investigational drug within 10 days before study entry.
* Uncontrolled infection at the time of enrollment.
* History of allogeneic transplantation.
* Manifestation of AML in the central nervous system.
* Pregnant or breast - feeding women.
* Men unable or unwilling to use adequate contraception methods from start of study treatment to minimum of six months after the last dose of chemotherapy.
* Women of childbearing potential except those who fulfill the following criteria: Post-menopausal or post-operative or continuous and correct application of a contraception method with a Pearl Index < 1 percent or sexual abstinence or vasectomy of the sexual partner.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | on day 56 after allogeneic SCT
  Disease-free survival

SECONDARY OUTCOMES:
Overall survival | 4 weeks, 8 weeks, and 24 weeks from randomization
  Overall survival
Rate of allogeneic transplantation | 4 weeks, 8 weeks, and 16 weeks from randomization
  Rate of allogeneic transplantation
Incidence of CR | at 4 weeks, 8 weeks, and 24 weeks from randomization
  Incidence of CR

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Schetelig, Prof Dr med, Study Chair — Universtitätsklinikum Dresden
Locations (18):
- Germany (18):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsmedizin Mannheim, Mannheim, Baden-Wurttemberg
  - Robert-Bosch-Krankenhaus, Stuttgart, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Rems-Murr-Kliniken gGmbH, Winnenden, Baden-Wurttemberg
  - Klinikum Augsburg, Augsburg, Bavaria
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Klinikum Nürnberg Nord, Nuremberg, Bavaria
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Universitätsklinikum Aachen, AÖR, Aachen, Nordrhein-Westphalen
  - Universitätsklinikum Essen (AöR), Essen, Nordrhein-Westphalen
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz, Rhineland-Palatinate
  - University Hospital, Dresden, Saxony
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Elblandkliniken Stiftung & Co. KG, Riesa, Saxony
  - Universitätsklinikum Halle (Saale), Halle, Saxony-Anhalt
  - Helios Klinikum Berlin Buch, Berlin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stelljes M, Middeke JM, Bug G, Wagner-Drouet EM, Muller LP, Schmid C, Krause SW, Bethge W, Jost E, Platzbecker U, Klein SA, Niederland J, Kaufmann M, Schafer-Eckart K, Baldauf H, Stolzel F, Trost S, Rollig C, von Bonin M, Egger-Heidrich K, Kunadt D, Steffen B, Hauptrock B, Schliemann C, Sockel K, Lang F, Kriege O, Schaffrath J, Reicherts C, Berdel WE, Serve H, Ehninger G, Schmidt AH, Mikesch JH, Bornhauser M, Schetelig J. Disease risk but not remission status determines transplant outcomes in AML: long-term outcomes of the ASAP trial. Blood. 2025 Nov 6;146(19):2293-2305. doi: 10.1182/blood.2025028730. PMID 40737595
- [Derived] Stelljes M, Middeke JM, Bug G, Wagner-Drouet EM, Muller LP, Schmid C, Krause SW, Bethge W, Jost E, Platzbecker U, Klein SA, Schubert J, Niederland J, Kaufmann M, Schafer-Eckart K, Schaich M, Baldauf H, Stolzel F, Petzold C, Rollig C, Alakel N, Steffen B, Hauptrock B, Schliemann C, Sockel K, Lang F, Kriege O, Schaffrath J, Reicherts C, Berdel WE, Serve H, Ehninger G, Schmidt AH, Bornhauser M, Mikesch JH, Schetelig J; Study Alliance Leukemia and the German Cooperative Transplant Study Group. Remission induction versus immediate allogeneic haematopoietic stem cell transplantation for patients with relapsed or poor responsive acute myeloid leukaemia (ASAP): a randomised, open-label, phase 3, non-inferiority trial. Lancet Haematol. 2024 May;11(5):e324-e335. doi: 10.1016/S2352-3026(24)00065-6. Epub 2024 Apr 4. PMID 38583455